CLINICAL TRIAL: NCT00658229
Title: Physical Exercise for Patients With Prostate Cancer During Androgen Deprivation Therapy - A Randomized Trial
Brief Title: The Physical Exercise and Prostate Cancer Study
Acronym: PEPC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Ullevaal University Hospital (Other); Norwegian School of Sport Sciences (Other); University of Alberta (Other); University of Oslo (Other); Norwegian Foundation for Health and Rehabilitation (Other); The Royal Norwegian Ministry of Health (Other)
Responsible Party: Principal Investigator, Lene Thorsen, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REK - 08/212b
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
Keywords: Exercise; Prostatic; Neoplasm; Androgen; Deprivation
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strength training group (Experimental): A four months strength training program during androgen deprivation therapy for prostate cancer patietns.
  Interventions: Behavioral: Strength training group
- Control group (No Intervention): Patients in the control group are not discouraged from performing normal activities. They are however asked not to start a strength training program or increase their activity level in the same period as the experimental group is performing their strength training program. We will offer the control group a modified strength training program after the post-intervention assessment.

INTERVENTIONS:
Behavioral: Strength training group — After 5-10 months on androgen deprivation therapy the patients in the intervention group go through a four months strength training intervention. The patients will perform three strength-training sessions per week, two under supervision of a sport instructor. Each session will consists of one-three sets of nine strength-training exercises, performed at an intensity of 6 or 10 repetitions of maximum (6-10 RM).
  Other Names: Exercise, Physical activity
  Arms: Strength training group

SUMMARY:
The purpose of this study is to determine the effectiveness of a four months strength training program on physical and psychological health in patients with prostate cancer during androgen deprivation therapy. It is hypothesized a beneficial effect of the intervention on physical and psychological health in patients with prostate cancer treated with androgen deprivation.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed locally advanced prostate cancer (clinical stage T2 and T3)
* Referred to RH and UUS for radiotherapy
* < 75 years
* Capable of reading and writing Norwegian
* Treating oncologist must approve of the subjects' participation
* Living within approximately 1 hour from Oslo by car or public transportation

Exclusion Criteria:

* Routinely resistance training with manuals
* Medication for osteoporosis (i.e. bisphosphonates)
* Conditions of a severity that contraindicate exercise without adjusted actions
* Mentally incompetent conditions
* Conditions of a severity that complicates the ability to participate in a supervised training program

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
lean body mass | before ADT, before and after the intervention

SECONDARY OUTCOMES:
bone mineral density, fat mass, body mass index, serological outcomes (including lipids, hormones and CRP), physical functioning, psycho-social functioning and muscle cellular outcomes (including muscle fiber size and function) | before ADT, before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lene Thorsen, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet- Radiumhospitalet HF, Montebello, Oslo County, Norway

REFERENCES:
- [Derived] Thorsen L, Nilsen TS, Raastad T, Courneya KS, Skovlund E, Fossa SD. A randomized controlled trial on the effectiveness of strength training on clinical and muscle cellular outcomes in patients with prostate cancer during androgen deprivation therapy: rationale and design. BMC Cancer. 2012 Mar 29;12:123. doi: 10.1186/1471-2407-12-123. PMID 22458865